CLINICAL TRIAL: NCT00002982
Title: A Phase II Trial of ICE Chemotherapy Followed by High Dose BEAM Chemotherapy With Autologous Peripheral Blood Progenitor Cell Transplantation in Patients >= 60 Years Old With Refractory or Relapsed Intermediate Grade Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Older Patients With Refractory or Relapsed Intermediate-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-004; CDR0000065505 (Registry Identifier: PDQ (Physician Data Query)); NCI-H97-1233
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic | interventions — Filgrastim; Carboplatin; Carmustine; Cytarabine; Etoposide; Ifosfamide; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: carmustine
Drug: cytarabine
Drug: etoposide
Drug: ifosfamide
Drug: melphalan
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with peripheral stem cell transplantation works in treating older patients with refractory or relapsed intermediate-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the efficacy and toxic effects of carmustine/etoposide/melphalan (ICE) chemotherapy followed by peripheral blood progenitor cell transplantation in patients with refractory or relapsed intermediate grade non-Hodgkin's lymphoma.
* Assess the ability of the ICE chemotherapy regimen, in conjunction with filgrastim, to mobilize peripheral blood stem cells.

OUTLINE: This is a descriptive pilot study.

Patients receive 3 cycles of induction chemotherapy with ifosfamide, carboplatin, and etoposide (ICE). Each cycle is given at least 14 days apart. Patients receive etoposide IV on days 1 through 3. Carboplatin and ifosfamide with mercaptoethane sulfonate is given IV over 24 hours on day 2.

During cycles 1 and 2, patients receive filgrastim (G-CSF) SC every 6 hours beginning on day 1 and continuing until the desired absolute neutrophil count (ANC) is attained.

Patients receive at least 24 hours of rest before PBPC infusion on day 0.

Following cycle 3, G-CSF is given SC beginning on day 6 and continuing until completion of PBPC collection. However, bone marrow will be harvested if an insufficient number of stem cells are collected after 5 leukaphereses.

Patients with residual disease limited to 2 sites receive radiation therapy twice a day within 2 weeks prior to high dose BEAM chemotherapy with carmustine, etoposide, cytarabine, and melphalan.

Patients receive carmustine IV on day -7. Etoposide and cytarabine are given IV every 12 hours on days -6 through -3. Melphalan is given IV on day -2.

G-CSF is administered every 12 hours beginning on day 1 and continuing until the desired ANC is attained. If ANC is attenuated on day 21, patients undergo a repeat bone marrow biopsy and receive filgrastim SC.

Patients are followed for 2 years posttransplant, then for 3 to 5 years at 4 month intervals and every 6 months following the fifth posttransplant.

PROJECTED ACCRUAL: This study will accrue 30 patients for the duration of 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Primary refractory intermediate grade non-Hodgkin's lymphoma (NHL) OR
* Untreated relapsed intermediate grade NHL with no more than 1 extranodal site of disease
* Biopsy proven relapse of diffuse large cell, diffuse mixed cell, diffuse small cleaved cell (excluding mantle cell lymphoma), follicular large cell, anaplastic large cell or immunoblastic NHL in recently attained complete response patients

PATIENT CHARACTERISTICS:

Age:

* 60 and over

Performance status:

* Karnofsky at least 80%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL unless there is a history of Gilbert's disease

Renal:

* No history of chronic renal insufficiency
* Creatinine no greater than 1.5 mg/dL or if greater than 1.5 mg/dL, then creatinine clearance must be at least 60 mL/min

Cardiovascular:

* No myocardial infarction within the past 6 months
* No unstable angina or cardiac arrhythmias other than chronic atrial fibrillation
* Normal cardiac function required; MUGA scan or stress ECG ejection fraction at least 50% without significant wall motion abnormalities

Pulmonary:

* Adequate pulmonary function defined as DLCO at least 50% of predicted value when corrected for patients hemoglobin and alveolar ventilation

Other:

* No medical illness unrelated to intermediate grade Non-Hodgkin's Lymphoma
* No uncontrolled infection
* No history of malignancy other than curatively treated cutaneous basal cell carcinoma; carcinoma in situ of the cervix; axillary node negative breast cancer without prior chemotherapy and disease free for more than 2 years; or prostate cancer with surgery alone and disease free for more than 2 years
* No lymphoblastic lymphoma, small noncleaved cell lymphoma, CNS lymphoma or CNS relapse of lymphoma
* Not HIV, HBV, and HCV positive

PRIOR CONCURRENT THERAPY:

* Concurrent enrollment in MSKCC protocol 96-17a allowed

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 2 prior chemotherapy regimens

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-01; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Treatment-related toxicity

SECONDARY OUTCOMES:
Efficacy in terms of 2-year disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States